CLINICAL TRIAL: NCT06119659
Title: Safety and Efficacy Clinical Study of Severe Hemophilia B Treatment With KL001
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Chief physician, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-KL001-001/01
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hemophilia B Without Inhibitor
MeSH Terms: interventions — KL001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KL001 injection solution (Experimental): Subjects will be dosed with three different dose of KL001 injection solution at 2.5x10^12 vg/kg to 1.0x10^13 vg/kg.
  Interventions: Drug: Low dose KL001; Drug: Middle dose KL001; Drug: High dose KL001

INTERVENTIONS:
Drug: Low dose KL001 — Subjects will be dosed with single dose of KL001 at 2.5x10^12 vg/kg.
  Other Names: rAAV vector
Drug: Middle dose KL001 — Subjects will be dosed with single dose of KL001 at 5.0x10^12 vg/kg.
  Other Names: rAAV vector
Drug: High dose KL001 — Subjects will be dosed with single dose of KL001 at 1.0x10^13 vg/kg.
  Other Names: rAAV vector

SUMMARY:
This is an open- label, non- randomized, uncontrolled, dose-escalation pilot study to evaluate the safety and efficacy of KL001 injection solution in hemophilia B subjects with ≤2 IU/dl residual FIX levels.

DETAILED DESCRIPTION:
This is an open- label, non- randomized, uncontrolled, dose-escalation pilot study to evaluate the safety and efficacy of KL001 injection solution in hemophilia B subjects with ≤2 IU/dl residual FIX levels. Nine subjects will be enrolled and administered with three different doses of KL001. Subjects will provide informed consent and then undergo screening assessments up to 1 month prior administration of KL001. All subjects will undergo 52 weeks safety observation and will be encouraged to enroll in an extension study to evaluate long- term safety of KL001 for a total 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥12 years of age.
2. Moderate/severe or severe hemophilia B (baseline FIX activity ≤2% of normal or documented history of FIX activity ≤2%).
3. At least 3 bleeding episodes per year that require on-demand treatment with FIX OR are treated with a prophylactic regimen of FIX.
4. At least 100 days exposure history to recombinant or plasma-derived FIX protein products.
5. No neutralizing antibodies to exogenous FIX protein products.
6. Willing and able to comply with study procedures and requirements.

Exclusion Criteria:

1. Suffering from chronic inflammatory muscle disease.
2. Positive in Hepatitis B or Hepatitis C.
3. Infection with HIV-1 or HIV-2 and CD4+T cell count ≤ 200/ μ L.
4. History of thrombosis or susceptibility to thrombosis.
5. Current or previous participation in another gene therapy study.
6. Has any other significant medical condition that the investigator feels would be a risk to the subject or would impede the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment- related adverse events | Infusion to the completion of study, about 52 weeks
  Number and severity of adverse events and serious adverse events and relationship to KL001
Antibody against KL001 AAV vector capsid protein | Infusion to the completion of study, about 52 weeks
  Immune response against AAV capsid will be evaluated by measurement of the total antibody and neutralizing antibody against AAV capsid protein in plasma samples collected at multiple timepoints after dosing up to 52 weeks
Factor IX inhibitor | Infusion to the completion of study, about 52 weeks
  Development of inhibitor against vector-derived Factor IX protein will be measured using bethesda method

SECONDARY OUTCOMES:
vector-derived FIX: C activity levels | From dosing day to week 52
  Peak and steady-state activity levels of vector-derived FIX: C
The annualized bleeding rate Before and After KL001 Infusion | From dosing day to week 52
  The annualized bleeding rate (ABR) will be calculated for all subjects through Week 52
The annualized use of FIX | From dosing day to week 52
  The use of on-demand FIX replacement therapy was recorded by dose (IU/kg) administered, and the annualized use of FIX replacement therapy was calculated for all subjects through Week 52.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD&MD, Principal Investigator — First Affiliated Hospital of Zhejiang University

IPD SHARING:
Plan to Share IPD: No